CLINICAL TRIAL: NCT03403413
Title: Cyclical Muscle Vibration in MS to Improve Walking
Brief Title: Muscle Vibration in MS to Improve Walking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ran out
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: F2177-P; RX002177 (Other: Louis Stokes VA Medical Center)
Record Dates: First submitted 2017-12-14; First posted 2018-01-18 (Actual); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Muscle Vibration (Experimental): Test feasibility of muscle vibration of tibialis anterior, rectus femoris, short head of biceps and tensor fasciae latae bilaterally during walking for 1 hour 3 times per week for 12 weeks to improve walking speed through improved coordination of hip, knee and ankle flexion.
  Interventions: Device: muscle vibration during walking

INTERVENTIONS:
Device: muscle vibration during walking — Baseline assessment of gait followed by 12 sessions (3/week for a month) of gait training with cyclic muscle vibration during walking emulating normal muscle activity of lower extremities in treatment group. Gait assessment both with and without muscle vibration were collected at follow-up after 12 sessions of gait training with muscle vibration.

SUMMARY:
The primary goal of this pilot study is to explore the feasibility of cyclic vibration (CV) of the lower extremity muscles to improve walking in individuals with gait deficits from multiple sclerosis (MS).

DETAILED DESCRIPTION:
This pilot study is designed to test the efficacy and safety of vibration at correcting the typical gait deficits that involve strength and coordination of multiple joints (hip, knee and ankle) in pre- and early swing phases of the gait cycle.

Aim 1: Develop a real-time control algorithm, timed by sensor detected gait events, to provide vibration emulating electromyographic (EMG) activity of target muscles during normal gait and verify its functionality in an able-body volunteer. Further, recruit 12 subjects (6 for CV and 6 controls) with gait deficits at the hip, knee and ankle from MS. Impose vibration during the gait cycle so that it emulates muscle activity pattern of normal gait. Perform baseline quantitative gait analyses to determine the spatio-temporal parameters, foot-to-floor clearance, kinematics, kinetics and patterns of EMG activity during walking with and without vibration in treatment group and without vibration in control group.

Aim 2: Implement 12 sessions (3/week for a month) of gait training with cyclic vibration emulating normal muscle activity of lower extremities in treatment group and gait training without vibration in control group and repeat baseline gait assessment to test the following hypotheses.

Hypothesis 1. Vibration of hip, knee and ankle muscles improves walking speed and foot-to-floor clearance through increased hip and knee pre-swing flexion and improved hip-knee coordination.

Hypothesis 2. Gait training with cyclic muscle vibration induces carryover effects that maintain improved walking after vibration is discontinued.

Hypothesis 3. Muscle vibration produces no untoward sensations or adverse physiological responses.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis reviewed and confirmed by neurologist per the revised McDonald criteria [ ]
* EDDS>3
* Age 18-70
* Fixed gait deficiency defined as being present for at least 3 months without improvement
* Hip, knee and ankle muscle weakness or increased extensor tone with difficulty to initiate a step
* Ability to ambulate at least 10ft with contact guard.
* Muscle vibration without untoward sensation.
* Sufficient upper extremity function to use walking aids (walkers, crutches, canes).
* Poor hip-knee-ankle coordination during swing
* Hip, knee and ankle joint range within normal limits.
* Ability to clearly understand written and oral direction in English to provide consent.
* BMI < 30
* Absence of psychological and cognitive problems or chemical dependency
* No acute orthopedic or medical complications

Exclusion Criteria:

* Presence of demand pacemakers.
* Edema of the affected limb/s.
* Uncontrolled seizures/epilepsy.
* Severe depression.
* Botulin toxin treatment within 12 months.
* Peripheral neuropathy.
* Respiratory disease.
* Chronic pain.
* Rapidly progressive course suggestive of Marburg variant, Hurst encephalomyelitis or PPMS with three or more system involvement.
* Concurrent treatment with Tysabri.
* Cardiac arrhythmias with associated hemodynamic instability.
* Lower extremity injuries that limit range of motion or function
* Joint problems (hip or leg) that limit range of motion or cause pain with movement
* Women during pregnancy
* Patients with a relapse in the 3 months prior to presentation for study evaluation
* Patients with more than two relapses within the past 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M. Selkirk, MD PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3
Pre-assignment Details: 3
Groups:
- Muscle Vibration: Test feasibility of muscle vibration of tibialis anterior, rectus femoris, short head of biceps and tensor fasciae latae bilaterally during walking for 1 hour 3 times per week for 12 weeks to improve walking speed through improved coordination of hip, knee and ankle flexion.
  Muscle vibration during walking: Baseline assessment of gait followed by 12 sessions (3/week for a month) of gait training with cyclic muscle vibration during walking emulating normal muscle activity of lower extremities and repeat gait assessment after gait training.
Period: Overall Study
Arm/Group | Muscle Vibration
Started (Case series of 3 subjects with multiple sclerosis.) | 5
Completed | 3
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Groups:
- Muscle Vibration: Test feasibility of muscle vibration of tibialis anterior, rectus femoris, short head of biceps and tensor fasciae latae bilaterally during walking for 1 hour 3 times per week for 12 weeks to improve walking speed through improved coordination of hip, knee and ankle flexion.
  muscle vibration during walking: Baseline assessment of gait followed by 12 sessions (3/week for a month) of gait training with cyclic muscle vibration during walking emulating normal muscle activity of lower extremities in treatment group and gait training without muscle vibration during walking in control group and repeat gait assessment after gait training.
Arm/Group | Muscle Vibration
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Kinematics of hip, knee and ankle flexion and speed and endurance of walking with and without vibration
  Participants
    United States | 3

OUTCOME MEASURES:

1. Primary Outcome: 10MWT
Description: speed (m/s)
Time Frame: baseline and after twelve 1 hour sessions in four weeks of gait training with muscle vibration. Outcome measures were tested both with and without muscle vibration and repeated measures were collected and averaged.
Population: Multiple sclerosis
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Subject A; Subject B; Subject C: Test feasibility of muscle vibration of tibialis anterior, rectus femoris, short head of biceps and tensor fasciae latae bilaterally during walking for 1 hour 3 times per week for 12 weeks to improve walking speed through improved coordination of hip, knee and ankle flexion.
  Muscle vibration during walking: Baseline assessment of gait followed by 12 sessions (3/week for a month) of gait training with cyclic muscle vibration during walking emulating normal muscle activity of lower extremities and repeat gait assessment after gait training.
Arm/Group | Subject A | Subject B | Subject C
Number analyzed (Participants) | 1 | 1 | 1
m/s
  Baseline | 1.1 (0) | 0.75 (0.09) | 1.39 (0.2)
  Follow-up without vibration | 1.295 (0.07) | 1.32 (0.009) | 2.18 (0.2)
  Follow-up with vibration | 1.39 (0.05) | 1.38 (0.05) | 1.86 (0.17)

2. Primary Outcome: Kinematics
Description: Peak hip, knee and ankle flexion during swing
Time Frame: baseline and after twelve 1 hour sessions in four weeks of gait training with muscle vibration. Repeated measures were collected and averaged
Population: Multiple sclerosis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Subject A | Subject B | Subject C
Number analyzed (Participants) | 1 | 1 | 1
degrees
  Volitional hip flexion pre-training | 24 (2.4) | 57 (7.4) | 27 (2.3)
  Volitional hip flexion post-vibration training | 38 (1.9) | 50 (5.8) | 30 (2.5)
  Volitional knee flexion pre-training | 49 (2.4) | 38 (16.3) | 72 (3.5)
  Volitional knee flexion post-vibration training | 61 (3.4) | 44 (15.8) | 74 (2.5)
  Volitional ankle dorsiflexion pre-training | 11 (2.7) | 13 (4.5) | 15 (4)
  Volitional ankle flexion post-vibration training | 14 (2.8) | 11 (3.2) | 15 (5.2)

3. Primary Outcome: Toe Clearance
Description: Toe clearance between foot and the ground during swing
Time Frame: as for outcome 2
Population: Multiple sclerosis
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Subject A | Subject B | Subject C
Number analyzed (Participants) | 1 | 1 | 1
mm
  Left leg volitional pre-training | 19.8 (4.4) | 30.6 (7.8) | 21.3 (3.5)
  Right Leg volitional pre-training | 17.6 (4.4) | 9.1 (2.5) | 21.5 (3.4)
  Left leg volitional post-vibration training | 30.2 (5.8) | 32 (5.8) | 25.5 (3.6)
  Right volitional post-vibration training | 25.4 (7.9) | 9.3 (3.6) | 24.7 (4.7)

4. Primary Outcome: Walking Distance
Description: Volitional walking distance at baseline and after gait training with vibration
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Subject A | Subject B | Subject C
Number analyzed (Participants) | 1 | 1 | 1
meters
  Volitional pre-training | 347 (0) | 252 (0) | 338 (0)
  Volitional post-vibration training | 361 (12) | 387 (11) | 406 (0)

ADVERSE EVENTS:
Time Frame: Data were collected over a period of 6 weeks from baseline to final evaluation
Groups:
- Feasibility: Test feasibility of muscle vibration of tibialis anterior, rectus femoris, short head of biceps and tensor fasciae latae bilaterally during walking for 1 hour 3 times per week for 12 weeks to improve walking speed through improved coordination of hip, knee and ankle flexion.
  Muscle vibration during walking: Baseline assessment of gait followed by 12 sessions (3/week for a month) of gait training with cyclic muscle vibration during walking emulating normal muscle activity of lower extremities and repeat gait assessment after gait training.
Arm/Group | Feasibility
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03403413/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT03403413/SAP_001.pdf